CLINICAL TRIAL: NCT05194215
Title: Real-world Observation of Medical Accuracy of a Novel AI-app
Acronym: ROMAN-AI
Status: Completed | Type: Observational
Sponsor: Ada Health GmbH (Industry)
Collaborators: Babes-Bolyai University (Other); Botnar Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: ROMAN-AI
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Gastrointestinal Issues; Respiratory Issues; Cardiovascular Issues; Genitourinary Issues; Musculoskeletal Issues; ENT Issues; Eye Issues; Neurologic Issues; Mental Health Issues

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ada WRA — The Ada WRA is a study-only device based on the Ada mobile app. The patient will use this device to answer questions regarding their symptoms but will not be given any feedback by the app.

SUMMARY:
This study aims to evaluate the performance of the suggestions made by the WRA by comparing Ada's list of suggested conditions and advice level to usual care and a gold-standard in a Romanian clinical setting.

DETAILED DESCRIPTION:
This pilot study investigates the performance of the Romanian version of Ada's Waiting Room Application in a clinical setting. The study will take place in a family doctor's practice in Cluj-Napoca, Romania. While waiting for their consultation with a family doctor, participants will complete an Ada assessment. The results of this assessment will not be available for viewing by the participants or the family practitioner. During and after consultation, the family practitioner will create two top 5 differential diagnoses list--one based on symptoms only and one based on physical examination and investigation results. The accuracy and comprehensiveness of Ada's differential diagnoses will be compared against the family practitioner's and a gold-standard.

ELIGIBILITY:
Inclusion Criteria:

* All patients under 60 years of age that enter the study sites and that are willing/able to provide consent will be included in the study, unless exclusion criteria are met.

Exclusion Criteria:

* Patients with severe injury/illness requiring immediate treatment
* Patients with traumatic injury
* Patients incapable of completing a health assessment (e.g. due to illiteracy, mental impairment or inebriation or other incapacity)
* Patients that are unfamiliar with mobile applications
* Patients that are seeking treatment for a chronic condition

Ages: 2 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The patients will be from the area of Cluj-Napoca, Romania and will be coming into their normal GP's office for a regular appointment.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Accuracy and comprehensiveness of the Ada WRA | about 5 months to gather the data
  Accuracy and comprehensiveness of the Ada WRA assessment evaluated against the gold standard differential diagnosis from the panel.

SECONDARY OUTCOMES:
Accuracy and comprehensiveness of the family practitioner | about 5 months to gather the data
  Accuracy and comprehensiveness of the family practitioner's differential diagnosis evaluated against the gold standard differential diagnosis from the panel.
Qualitative data on the chronology usability, usefulness and acceptance | about 3 months to gather the data
  Gathered from surveys from patient, study nurse, and doctor

CONTACTS AND LOCATIONS:
Overall Officials: Marius-Ionuț Ungureanu, MD, PhD, Principal Investigator — Cluj School of Public Health; Madalina A Coman, PhD, Principal Investigator — Cluj School of Public Health
Locations (1):
- Dr. Claudia Pîrșan, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared if there is a reasonable request and this request is approved by the IRB in charge of the study.